CLINICAL TRIAL: NCT01195532
Title: An Open-randomized, Balanced, Crossover Bioequivalence Study to Compare One MR Tablet of 60 mg Gliclazide and Two MR Tablets of 30 mg Gliclazide in Healthy Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsingjin E. Liu, MD, PhD., Taipei Medical University WanFang Hospital
Other Study IDs: A29GLI60-1; E814A29E11; E814A29E11 (Other: Rosetta)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Hyperglycemia; Diabetes
Keywords: hypoglycemic drug
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Crossover
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gliclazide/2: 60 mg*1 for T 30 mg*2 For R
- Reference and test drug: Reference: 30 mg *2 Test: 60 mg *1

SUMMARY:
The 2 × 2 crossover designed study is to evaluate the bioequivalence of two different MR tablets of gliclazide after single oral administration at the same doses to healthy subjects.

DETAILED DESCRIPTION:
The 2 × 2 crossover designed study is to evaluate the bioequivalence of two different MR tablets of gliclazide after single oral administration at the same doses to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled into the study according to the following criteria:

1. Subjects must be male at the age of 20-40 years old in good health on the basis of medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.
2. Vital signs (after 3 minutes resting in a upright position) which are within the following ranges:

   Ear body temperature between 35.0-37.5 °C. Systolic blood pressure, 90-140 mm Hg. Diastolic blood pressure, 50-90 mm Hg. Pulse rate, 50-90 bpm. Fasting blood glucose, < 100 mg/dL.
3. Body weight must be greater than 50 kg and within -20 to +20% of ideal body weight.
4. Able to sign informed consent prior to study.
5. Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

Subjects meet any of the following criteria during pre-study examination evaluation will be excluded from entry into or continuation in the study:

1. Use of any prescription medication within 14 days prior to dosing.
2. Use of over-the-counter medications or vitamins within 14 days prior to dosing.
3. Significant illness within 2 weeks prior to dosing.
4. Participation in any clinical investigation within 2 months prior to dosing or longer than required by local regulation.
5. Donate or loss more than 500 mL of blood within 3 months prior to dosing.
6. Presence of cardiovascular disease.
7. Presence of gastrointestinal disease.
8. Presence of asthma or lung disease.
9. Presence of liver disease, hepatitis B, hepatitis C or liver injury as indicated by an abnormal liver function profile such as GOT, GPT,gama-GT, alkaline phosphatase, serum bilirubin, HBsAg, or Anti-HCV.
10. Presence of impaired renal function as indicated by abnormal creatinine or BUN values or abnormal urinary constituents (e.g., albuminuria).
11. Presence of neurological disease.
12. Presence of psychiatrical disease.
13. Subject is known for HIV infected.
14. A known hypersensitivity to gliclazide or its analogs.
15. History of drug or alcohol abuse within 12 months prior to dosing.
16. Permanent confinement to an institution.
17. Individuals are judged by the investigator or pharmacokineticist to be undesirable as subjects for other reasons.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health subjects
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
AUC0-t, AUC0-∞, Cmax, Tmax, T1/2, and MRT in plasma will be determined with gliclazide concentrations by non-compartment methods. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Hsingjin E Liu, MD, PhD E Liu, MD, PhD, Principal Investigator — Taipei Medical University - Municipal Wan Fang Hospital
Locations (1):
- Taipei Medical University - Municipal Wan Fang Hospital, Taipei, Taiwan, Taiwan